CLINICAL TRIAL: NCT04949373
Title: Evaluation of the Efficacy of High Intensity Laser (HILT) Therapy in Idiopathic Carpal Tunnel Syndrome
Brief Title: High Intensity Laser Therapy in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Selma Eroğlu, Principal Investigator / Medical Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Afyonkarahisar Health Sciences
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Carpal Tunnel Syndrome; Entrapment Neuropathy; Median Neuropathy; Musculoskeletal Diseases
Keywords: Carpal Tunnel Syndrome; Median Neuropathy; High intensity laser therapy; Nerve conduction studies; Hand function
MeSH Terms: conditions — Carpal Tunnel Syndrome; Charcot-Marie-Tooth Disease; Median Neuropathy; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT+nerve/tendon gliding exercise+rest splint (Experimental): Patients will receive pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for three weeks (one session per day for a total of 15 sessions). A 3-phase treatment program will be performed in each session, and a physiotherapist will then apply nerve/tendon gliding exercises program to the patients once daily. The patients will use rest splint at night.
  Interventions: Device: High-intensity laser therapy (HILT)
- Sham HILT+nerve/tendon gliding exercise+rest splint (Sham Comparator): Patients will receive sham laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for three weeks (one session per day for a total of 15 sessions). A 3-phase treatment program will be performed in each session, and a physiotherapist will then apply nerve/tendon gliding exercises program to the patients once daily . The patients will use rest splint at night.
  Interventions: Device: Sham High-intensity laser therapy (sham HILT)

INTERVENTIONS:
Device: High-intensity laser therapy (HILT) — High intensity laser therapy-Patients will receive pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of three weeks, and one session per day for a total of 15 sessions. A 3-phase treatment program will be performed on each session.
  Other: Tendon and nerve gliding exercises will be performed three times a day with 10 repetitions each time for 3 weeks. Exercises will be performed by a trained physiotherapist.
  Other: Rest splint(at night) Participants will be splinted in neutral position with standard cotton-polyester splints.The patients will be encouraged to use the splints during nighttime for 12 weeks.
  Arms: HILT+nerve/tendon gliding exercise+rest splint
Device: Sham High-intensity laser therapy (sham HILT) — Sham high intensity laser therapy-Participants will receive pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of three weeks, and one session per day for a total of 15 sessions.
  Other: Tendon and nerve gliding exercises will be performed three times a day with 10 repetitions each time for 3 weeks. Exercises will be performed by a trained physiotherapist.
  Other: Rest splint(at night) Participants will be splinted in neutral position with standard cotton-polyester splints.The patients will be encouraged to use the splints during nighttime for 12 weeks.
  Arms: Sham HILT+nerve/tendon gliding exercise+rest splint

SUMMARY:
This research aims to investigate the effect of high-intensity laser therapy on pain, function, nerve conduction studies and grip strength in patients with idiopathic carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy, and it causes numbness and tingling in the hand, atrophy and muscle weakness in the later stages. Any condition that increases the volume of the carpal tunnel and narrows the diameter of the tunnel may increase the compression of the median nerve under the transverse carpal ligament and cause symptoms. In majority of cases, no cause can be found and it is called "idiopathic".

While the diagnosis of CTS is made by the patient's history and physical examination methods, the diagnosis is confirmed with use of electrophysiological examination. Physical therapy, non-steroidal anti-inflammatory drug use, local steroid injection, hand-wrist rest splint, nerve/tendon gliding exercises; Physiotherapy modalities such as therapeutic ultrasound and laser are among the conservative treatment methods of CTS. Despite the effectiveness of surgery in the treatment of severe CTS cases, as is known, surgical treatment is not without risk. Therefore, mild to moderate CTS is treated conservatively.

Laser therapy is one of the physical therapy modalities, low-intensity laser therapy (LILT), whose biological effects occur secondary to direct photochemical effect and are not the result of thermal effects. High-intensity laser therapy (HILT), which has been widely used recently, is frequently used since it has small and slow light absorption from chromophores. HILT is not a concentrated light, but it diffuses in all directions (scattering phenomenon). This supports the wider effectiveness of HILT. HILT also has effects such as increased mitochondrial oxidative reactions, increased production of adenosine triphosphate, RNA and DNA (photochemical effect), increased tissue stimulation (photobiological), and reduced pain and inflammation. HILT, which has recently found many uses in musculoskeletal diseases, can affect a wider and deeper area in the tissues compared to the widely used LILT. Although there are many studies on the effectiveness of LILT therapy in CTS, there are few trials to study the effectiveness of HILT on clinical and electrophysiological parameters in CTS.

This investigation is designed as double-blind prospective sham controlled randomized study.

Participants were randomized into 2 groups: 1) HILT + nerve/tendon gliding exercises + rest splint and 2) Sham HILT+ nerve/tendon gliding exercises + rest splint

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate idiopathic carpal tunnel syndrome (clinically diagnosed and electrophysiologically confirmed CTS)

Exclusion Criteria:

* Diabetes mellitus,hypothyroidism, rheumatic diseases, acromegaly
* Polyneuropathy,
* Ipsilateral brachial plexopathy and traumatic nerve injury of the upper extremity
* Previous injection into the carpal tunnel and physical therapy within in the preceding 6 months
* Pregnancy
* History of malignancy
* Patients with cochlear implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
The Boston carpal tunnel questionnaire: 0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  This questionnaire determines CTS-specific symptom severity and functional outcome using a scale for each. Symptom severity subgroup is determined using 11 questions scored from 1 to 5 and one can get 55 points at most. The higher the score, the higher the symptom severity. The function subgroup questions the difficulty of 8 functional activities scored from 1 to 5 and one can get 40 points at most. The higher the score, the worse the functional capacity.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) [ Time Frame: 0(Baseline), Change from Baseline VAS at 3rd and 12th weeks ] | 0(Baseline) and at 3rd and 12th weeks
  Pain intensity will be measured with visual analogue scale (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.
Median nerve distal motor latency.Time Frame: 0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  The compound muscle action potential amplitude(CMAP) will be obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode will be placed on the muscle belly and the reference electrode will be placed on the tendon insertion. The median nerve will be stimulated 8 cm proximal to the active recording electrode. Distal motor latencies will be measured from the onset of stimulus artifact to the onset of the CMAP.
Sensory nerve conduction velocity Time Frame: 0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  Sensory nerve action potential amplitudes (SNAP) will be obtained using an orthodromic method and recorded by surface electrodes placed at the wrist The median nerves will be stimulated at the proximal and distal interphalangeal joints of the index finger . Distal sensory latencies will be measured from the onset of the stimulus artifact to the onset of the SNAP. Sensory nerve conduction velocity will be calculated dividing the distance by the distal sensory latency.
Median nerve compound muscle action potential amplitude (CMAP): Time Frame: 0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  The CMAPs will be obtained via surface electrodes placed on the abductor pollicis brevis muscle. The active recording electrode will be placed on the muscle belly, and the reference electrode will be placed on the tendon insertion. The median nerve will be stimulated 8 cm proximal to the active recording electrode. The amplitude of CMAP will be measured from baseline to negative peak.
Median sensory nerve action potential amplitudes: Time Frame: 0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  Sensory nerve action potential amplitudes (SNAP) will be obtained using an orthodromic method and recorded by surface electrodes placed at the wrist The median nerves will be stimulated at the proximal and distal interphalangeal joints of the index finger and palm . Distal sensory latencies will be measured from the onset of the stimulus artifact to the onset of the SNAP.
Grip strength: Time Frame:0(Baseline), Change from Baseline at 3rd and 12th weeks | 0(Baseline) and at 3rd and 12th weeks
  In the evaluation of grip strength, a hand dynamometer (JAMAR) will be used for grip strength and a pinchmeter will be used for the evaluation of the pulp to pulp grip. The patient will perform three consecutive tests while sitting with their shoulder abducted and neutrally rotated, elbow flexed at 90°, and forearm and wrist in neutral position.The best of these measurements will be recorded in kilograms.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Merkez, Afyonkarahi̇sar, Turkey (Türkiye)

REFERENCES:
- [Background] Bekhet AH, Ragab B, Abushouk AI, Elgebaly A, Ali OI. Efficacy of low-level laser therapy in carpal tunnel syndrome management: a systematic review and meta-analysis. Lasers Med Sci. 2017 Aug;32(6):1439-1448. doi: 10.1007/s10103-017-2234-6. Epub 2017 Jun 5. PMID 28580494
- [Background] Dundar U, Turkmen U, Toktas H, Ulasli AM, Solak O. Effectiveness of high-intensity laser therapy and splinting in lateral epicondylitis; a prospective, randomized, controlled study. Lasers Med Sci. 2015 Apr;30(3):1097-107. doi: 10.1007/s10103-015-1716-7. Epub 2015 Jan 23. PMID 25614134
- [Background] Guner A, Altan L, Kasapoglu Aksoy M. The effectiveness of the low-power laser and kinesiotaping in the treatment of carpal tunnel syndrome, a pilot study. Rheumatol Int. 2018 May;38(5):895-904. doi: 10.1007/s00296-018-4020-6. Epub 2018 Mar 28. PMID 29594333
- [Background] Ezzati K, Laakso EL, Salari A, Hasannejad A, Fekrazad R, Aris A. The Beneficial Effects of High-Intensity Laser Therapy and Co-Interventions on Musculoskeletal Pain Management: A Systematic Review. J Lasers Med Sci. 2020 Winter;11(1):81-90. doi: 10.15171/jlms.2020.14. Epub 2020 Jan 18. PMID 32099632
- [Background] Yagci I, Elmas O, Akcan E, Ustun I, Gunduz OH, Guven Z. Comparison of splinting and splinting plus low-level laser therapy in idiopathic carpal tunnel syndrome. Clin Rheumatol. 2009 Sep;28(9):1059-65. doi: 10.1007/s10067-009-1213-0. Epub 2009 Jun 21. PMID 19544043